CLINICAL TRIAL: NCT03537963
Title: Developing and Testing an mHealth Stepped-Care Intervention for Sleep Disturbance in HCT Survivors
Brief Title: Improving Sleep in BMT Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-19486
Record Dates: First submitted 2018-05-09; First posted 2018-05-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sleep Disturbance; Sleep Disorder
Keywords: HCT survivors; hematopoietic stem cell transplant (HCT); survivors of hematopoietic stem cell transplant
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Intervention Model Description: After the first part of the study (Qualitative Interviews), the hematopoietic cell transplant (HCT) survivors will be randomized to 3 different study arms for the intervention portion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-Intervention Qualitative Interviews (Other): Hematopoietic cell transplant (HCT) survivors, caregivers and clinicians will participate in this part of the study. HCT survivor participants will be asked to nominate and provide contact information for the person who was their primary caregiver before, during, or after their HCT hospitalization. All participants will be asked to participate in either an in-person or telephone interview that will last approximately 1 hour. The interview will be digitally audio-recorded and will ask questions on the trajectory of sleep disturbance in HCT recipients and strategies to manage common barriers to quality sleep, as well as discuss the planned intervention for sleep disturbance in HCT survivors.
  Interventions: Other: Qualitative Interviews
- mHealth Stepped-care Intervention (Experimental): For HCT survivors randomized to this group: Baseline survey, followed by mHealth Stepped-care intervention, post-intervention questionnaire and interview.
  Interventions: Other: mHealth Stepped-care Intervention; Other: Questionnaire; Other: Interview
- Educational Control Condition (Active Comparator): For HCT survivors randomized to this group: Baseline survey, followed by Educational Control intervention, post-intervention questionnaire and interview.
  Interventions: Other: Educational Control Condition; Other: Questionnaire; Other: Interview
- mHealth Stepped-care Intervention + virtual reality relaxation (Experimental): For HCT survivors randomized to this group: Baseline survey, followed by mHealth Stepped-care intervention + virtual reality relaxation component, post-intervention questionnaire and interview.
  Interventions: Other: mHealth Stepped-care Intervention; Other: Questionnaire; Other: Interview; Other: Virtual Reality

INTERVENTIONS:
Other: mHealth Stepped-care Intervention — Test of the feasibility and acceptability of an mHealth stepped-care intervention for sleep disturbance in HCT survivors, to compare with the control group.
  Arms: mHealth Stepped-care Intervention; mHealth Stepped-care Intervention + virtual reality relaxation
Other: Educational Control Condition — General health education for cancer survivors provided in NCI booklets entitled Facing Forward: Life After Cancer Treatment and Coping With Advanced Cancer.
  Arms: Educational Control Condition
Other: Questionnaire — After the intervention, participants will be asked to complete a questionnaire to provide feedback on the intervention.
  Arms: Educational Control Condition; mHealth Stepped-care Intervention; mHealth Stepped-care Intervention + virtual reality relaxation
Other: Interview — Qualitative interviews will be gathered after the participants have completed participation in the new intervention to gather data to inform future refinements of the intervention.
  Arms: Educational Control Condition; mHealth Stepped-care Intervention; mHealth Stepped-care Intervention + virtual reality relaxation
Other: Qualitative Interviews — To conduct qualitative interviews with patients, caregivers, and clinicians regarding sleep disturbance in HCT survivors and on preferences for a new mHealth intervention for sleep disturbance. Separate panels of 10 HCT survivors, 10 caregivers who were the primary caregiver of an HCT survivor during or after the inpatient HCT hospitalization, and 5-10 HCT clinicians will be recruited for individual qualitative interviews via telephone or in person.
  Other Names: Questionnaire
  Arms: Pre-Intervention Qualitative Interviews
Other: Virtual Reality — The intervention will comprise six 360º videos of relaxing natural landscapes from which patients can choose (i.e., beaches, tropical scenes, calm thunderstorms, snowfall). Participants will also choose an audio accompaniment: a progressive muscle relaxation script, a deep breathing exercise script, a mindfulness meditation script, or scene-relevant audio (e.g., waves crashing for the beach scene).
  Other Names: VR
  Arms: mHealth Stepped-care Intervention + virtual reality relaxation

SUMMARY:
The purpose of this study is to:

To test a new intervention for sleep disturbance among hematopoietic cell transplant survivors. About 60 hematopoietic cell transplant (HCT) survivors will participate in this intervention.

Preliminary Steps: To conduct qualitative interviews with patients, caregivers, and clinicians regarding sleep disturbance in hematopoietic cell transplant (HCT) survivors and on preferences for a new mHealth intervention for sleep disturbance. About 30 individuals (10 HCT survivors, 10 caregivers and 5-10 clinicians) will participate in this part of the study.

DETAILED DESCRIPTION:
Investigators will collect qualitative interview data from HCT survivors, caregivers, and clinicians to inform the development of a new mHealth intervention. Then, this new intervention will be developed by adapting existing interventions that were originally designed for other cancer and non-cancer populations.A virtual reality relaxation component will also be developed as an adjunct to the mHealth stepped-care intervention.

Intervention participants will complete a baseline survey via the internet about their demographics, health, and well-being. The baseline survey also includes questions about their sleep and will take approximately 1 hour to complete.

Participants will then be provided brief behavioral therapy through the mHealth intervention. Participants would be monitored passively via actigraphy for the next 30 days. Those who continue demonstrating clinically significant sleep disturbance 30 days after starting the intervention would then receive a more intensive therapy with a trained therapist via videoconferencing. This videoconferencing therapy, adapted from cognitive behavioral therapy for insomnia, will also be a built-in part of the mHealth intervention. Thus, the new mHealth intervention will be delivered via mobile device to enhance disseminability and improve access for survivors who typically live long distances from their HCT center.

Then Sixty HCT survivors with clinically significant sleep disturbance will be recruited 90 days after HCT and be block-randomized based on sex to receive usual care (n=20), the new mHealth stepped-care intervention (n=20), or the new mHealth stepped-care intervention +virtual relaxation component (n=20). Outcomes will be assessed before randomization as well as 30 and 60 days later. Participants will complete a validated self-report measure of sleep disturbance, and for objective measurement of sleep participants will be asked to wear a Fitbit and allow Fitbit data to be uploaded to the intervention for customizing individuals' interventions.

After the intervention, participants will be asked to complete a questionnaire to provide feedback on the intervention and participate in a post-intervention interview with a member of the study team.

ELIGIBILITY:
Inclusion Criteria:

FOR QUALITATIVE INTERVIEWS PRE-TEST

* HCT survivors: Potentially eligible patients will be approached in person during a routine outpatient appointment at Moffitt Cancer Center or via telephone.
* Additional eligibility criteria for HCT survivors will require that participants have undergone an allogeneic HCT within the previous 6 months - 2 years for a hematologic malignancy and be reporting clinically significant sleep disturbance (≥ 4 on a scale of 0 - 10).
* Caregivers of HCT survivors: Patient participants will be asked to nominate and provide contact information for the person who was their primary caregiver before, during, or after their HCT hospitalization.
* Adults ≥ 18 years old
* Able to speak and read English
* Able to provide informed consent
* Have no documented or observable severe and untreated neurological or psychiatric disorders that would preclude participation (e.g., psychosis).
* Clinicians: Eligible clinicians will be oncologists, nurses, or other clinicians at the Moffitt Cancer Center Blood and Marrow Transplant Program.

FOR INTERVENTION GROUPS

* Are ≥18 years of age
* Have been diagnosed with a hematologic malignancy
* Were discharged after allogeneic HCT within the previous 110 days (to allow for those who return to clinic within approximately 2 weeks of their planned 90-day clinic visit)
* Are experiencing clinically significant sleep disturbance
* Have never been diagnosed with nor are at high risk of sleep disorders that are unlikely to be ameliorated with behavioral treatment (e.g., obstructive sleep apnea, restless leg syndrome) as assessed using the Duke Structured Interview for Sleep Disorders
* Are able to sign informed consent
* Do not have any untreated or severe psychiatric or neurological disorders or other disabilities that would impair their ability to participate in this study.

Exclusion Criteria:

* Do not meet Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Rate of Participant Completion of Study | Up to 60 days
  The study will be considered feasible if 70% of those who participate complete the intervention.
Rate of Participant Satisfaction | 60 days post intervention
  The study will be considered acceptable if 50% of eligible patients approached for study participation sign consent and if > 50% of the mHealth stepped-care intervention group participants report that they are at least "mostly satisfied" with the intervention on a validated satisfaction scale. That is, at least half report an average score of ≥ 3 on a scale of 1 to 4 on this instrument.

SECONDARY OUTCOMES:
Rate of Sleep Disturbance | 60 days post intervention
  Sleep disturbance will be operationalized by scores on the Pittsburgh Sleep Quality Index and sleep efficiency (the percentage of time spent in bed that is spent asleep). For secondary efficacy analyses participants will be categorized as having sleep disturbance if their Pittsburgh Sleep Quality Index score is ≥ 5 (for subjectively-measured sleep disturbance) and if their sleep efficiency is <85% (for objectively-measured sleep disturbance).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Gonzalez, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided